CLINICAL TRIAL: NCT01949649
Title: Dissonance Eating Disorder Prevention: Clinician Led, Peer Led vs Web Delivered (Formerly: Effectiveness Trial of Peer-Led Dissonance Eating Disorder Prevention Groups)
Brief Title: Dissonance Eating Disorder Prevention: Clinician Led, Peer Led vs Web Delivered
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MH097720
Record Dates: First submitted 2013-09-17; First posted 2013-09-24 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Eating Disorder Prevention
Keywords: body image; body dissatisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Peer-Led Group Intervention (Active Comparator): In the Peer-Led Group Intervention, participants voluntarily engage in verbal, written, and behavioral exercises in which they critique the thin-ideal ideal during 4 1-hr sessions and in homework activities which are led by peer leaders.
  Interventions: Behavioral: Peer-Led Group Intervention
- Clinician-Led Group Intervention (Active Comparator): In the Clinician-Led Group Intervention, participants voluntarily engage in verbal, written, and behavioral exercises in which they critique the thin-ideal ideal during 4 1-hr sessions and in homework activities which are led by University clinicians.
  Interventions: Behavioral: Clinician-Led Group Intervention
- Internet-Based Intervention (Active Comparator): The Internet-Based Intervention consists of 6 40-min modules involving user-driven self-education activities and games (e.g., role-plays), writing/video contests, and off-line exercises designed to induce dissonance regarding pursuit of the thin-ideal, mirroring activities from the group Body Project.
  Interventions: Behavioral: Internet-Based Intervention
- Education Video (Active Comparator): The Education Video describes eating disorders, their adverse effects, and the need for treatment, which is key information to provide to young women at elevated risk for eating disorders due to body dissatisfaction.
  Interventions: Behavioral: Education Video

INTERVENTIONS:
Behavioral: Peer-Led Group Intervention
  Arms: Peer-Led Group Intervention
Behavioral: Internet-Based Intervention
  Arms: Internet-Based Intervention
Behavioral: Clinician-Led Group Intervention
  Arms: Clinician-Led Group Intervention
Behavioral: Education Video
  Arms: Education Video

SUMMARY:
Five percent of young women meet criteria for anorexia nervosa, bulimia nervosa, or binge eating disorder, with another 5% meeting criteria for Eating Disorder Not Otherwise Specified (ED-NOS), which includes subthreshold variants of these disorders. Over half of those presenting for eating disorder treatment meet criteria for ED-NOS and both threshold cases and ED-NOS are marked by chronicity, relapse, distress, functional impairment, and increased risk for future obesity, depression, suicide attempts, anxiety disorders, substance abuse, morbidity, and mortality. Anorexia and bulimia nervosa show stronger relations to suicide attempts, outpatient/inpatient treatment, and functional impairment than most other psychiatric disorders. Treatment of eating disorders is very expensive, similar to the cost for schizophrenia treatment, and is effective for only 40-60% of patients. Thus, a public health priority is to develop and disseminate effective eating disorder prevention programs.

DETAILED DESCRIPTION:
Although dozens of eating disorder prevention programs have been evaluated, only a dissonance-based program (the Body Project) has significantly reduced future onset of threshold and subthreshold eating disorders through long-term follow-up. An effectiveness trial found that the Body Project produced significant reductions in risk factors, eating disorder symptoms, and functional impairment relative to educational brochure controls, with some effects persisting through 3-yr follow-up when high school clinicians recruited students and delivered the program. These trials confirm the efficacy and effectiveness of the Body Project, but revealed a key dissemination barrier; it can be difficult to identify and recruit clinicians at high schools and colleges with the time and expertise to competently deliver the program.

One solution to this key dissemination barrier is to train students in established peer leader programs at colleges to recruit high-risk students and deliver the program. Another solution to this dissemination barrier would be to deliver the Body Project via the Internet.

Because peer-led groups and Internet delivery of the Body Project could markedly extend the reach and sustainability of this evidence-based program, we propose to conduct the first large multi-site effectiveness trial that directly compares the effects and cost effectiveness of peer-led Body Project groups, the eBody Project intervention, and clinician-led Body Project groups to an educational video control condition.

ELIGIBILITY:
Inclusion Criteria:

* Body image concerns
* Attend University of Oregon, Oregon State University, University of Texas at Austin, or Southwestern University

Exclusion Criteria:

* Meeting criteria for anorexia nervosa, bulimia nervosa, or binge eating disorder
* Suicidal ideation

Ages: 17 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 680 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change over time: Eating disorder diagnostic interview | baseline obtained on intake, 1 month post intervention and at 6mo, 1-, 2-, and 3-year follow-ups
  Participants will complete an interview assessing Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) eating disorder symptoms.

SECONDARY OUTCOMES:
Change over time: Thin-ideal internalization | baseline obtained on intake, 1 month post intervention and 6mo-, 1-, 2-, & 3-year followups
  Thin-ideal internalization will be assessed with the 8-item Ideal-Body Stereotype Scale-Revised. Participants respond using a 5-point response format.

OTHER OUTCOMES:
Change over time: Body Dissatisfaction | baseline obtained on intake, 1 month post intervention and at 6mo, 1-, 2- & 3-yr followups
  Body dissatisfaction will be assessed with the Body Dissatisfaction Scale. Respondents rate their level of satisfaction with 9 body parts on 6-point scales.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, PhD, Principal Investigator — Oregon Research Institute
Locations (3):
- United States (3):
  - Oregon Research Institute, Corvallis, Oregon
  - Oregon Research Institute, Eugene, Oregon
  - University of Texas at Austin, Austin, Texas

REFERENCES:
- [Background] Stice E, Rohde P, Gau J, Shaw H. An effectiveness trial of a dissonance-based eating disorder prevention program for high-risk adolescent girls. J Consult Clin Psychol. 2009 Oct;77(5):825-34. doi: 10.1037/a0016132. PMID 19803563
- [Background] Stice E, Rohde P, Shaw H, Gau J. An effectiveness trial of a selected dissonance-based eating disorder prevention program for female high school students: Long-term effects. J Consult Clin Psychol. 2011 Aug;79(4):500-8. doi: 10.1037/a0024351. PMID 21707136
- [Background] Stice E, Rohde P, Shaw H, Marti CN. Efficacy trial of a selective prevention program targeting both eating disorder symptoms and unhealthy weight gain among female college students. J Consult Clin Psychol. 2012 Feb;80(1):164-170. doi: 10.1037/a0026484. Epub 2011 Nov 28. PMID 22122289
- [Background] Stice E, Rohde P, Durant S, Shaw H. A preliminary trial of a prototype Internet dissonance-based eating disorder prevention program for young women with body image concerns. J Consult Clin Psychol. 2012 Oct;80(5):907-16. doi: 10.1037/a0028016. Epub 2012 Apr 16. PMID 22506791
- [Background] Hudson JI, Hiripi E, Pope HG Jr, Kessler RC. The prevalence and correlates of eating disorders in the National Comorbidity Survey Replication. Biol Psychiatry. 2007 Feb 1;61(3):348-58. doi: 10.1016/j.biopsych.2006.03.040. Epub 2006 Jul 3. PMID 16815322
- [Background] Stice E, Marti CN, Rohde P. Prevalence, incidence, impairment, and course of the proposed DSM-5 eating disorder diagnoses in an 8-year prospective community study of young women. J Abnorm Psychol. 2013 May;122(2):445-57. doi: 10.1037/a0030679. Epub 2012 Nov 12. PMID 23148784
- [Background] Wade TD, Bergin JL, Tiggemann M, Bulik CM, Fairburn CG. Prevalence and long-term course of lifetime eating disorders in an adult Australian twin cohort. Aust N Z J Psychiatry. 2006 Feb;40(2):121-8. doi: 10.1080/j.1440-1614.2006.01758.x. PMID 16476129
- [Background] Fairburn CG, Harrison PJ. Eating disorders. Lancet. 2003 Feb 1;361(9355):407-16. doi: 10.1016/S0140-6736(03)12378-1. PMID 12573387
- [Background] Crow SJ, Peterson CB, Swanson SA, Raymond NC, Specker S, Eckert ED, Mitchell JE. Increased mortality in bulimia nervosa and other eating disorders. Am J Psychiatry. 2009 Dec;166(12):1342-6. doi: 10.1176/appi.ajp.2009.09020247. Epub 2009 Oct 15. PMID 19833789
- [Background] le Grange D, Binford RB, Peterson CB, Crow SJ, Crosby RD, Klein MH, Bardone-Cone AM, Joiner TE, Mitchell JE, Wonderlich SA. DSM-IV threshold versus subthreshold bulimia nervosa. Int J Eat Disord. 2006 Sep;39(6):462-7. doi: 10.1002/eat.20304. PMID 16715488
- [Background] Schmidt U, Lee S, Perkins S, Eisler I, Treasure J, Beecham J, Berelowitz M, Dodge L, Frost S, Jenkins M, Johnson-Sabine E, Keville S, Murphy R, Robinson P, Winn S, Yi I. Do adolescents with eating disorder not otherwise specified or full-syndrome bulimia nervosa differ in clinical severity, comorbidity, risk factors, treatment outcome or cost? Int J Eat Disord. 2008 Sep;41(6):498-504. doi: 10.1002/eat.20533. PMID 18433024
- [Background] Newman DL, Moffitt TE, Caspi A, Magdol L, Silva PA, Stanton WR. Psychiatric disorder in a birth cohort of young adults: prevalence, comorbidity, clinical significance, and new case incidence from ages 11 to 21. J Consult Clin Psychol. 1996 Jun;64(3):552-62. PMID 8698949
- [Background] Striegel-Moore RH, Leslie D, Petrill SA, Garvin V, Rosenheck RA. One-year use and cost of inpatient and outpatient services among female and male patients with an eating disorder: evidence from a national database of health insurance claims. Int J Eat Disord. 2000 May;27(4):381-9. doi: 10.1002/(sici)1098-108x(200005)27:43.0.co;2-u. PMID 10744844
- [Background] Stice E, Shaw H, Burton E, Wade E. Dissonance and healthy weight eating disorder prevention programs: a randomized efficacy trial. J Consult Clin Psychol. 2006 Apr;74(2):263-75. doi: 10.1037/0022-006X.74.2.263. PMID 16649871
- [Derived] Stice E, Desjardins C, Shaw H, Siegel S, Gee K, Rohde P. Prevalence, incidence, impairment, course, and diagnostic progression and transition of eating disorders, overweight, and obesity in a large prospective study of high-risk young women. J Psychopathol Clin Sci. 2025 May;134(4):427-437. doi: 10.1037/abn0000965. Epub 2024 Nov 7. PMID 39509183
- [Derived] Stice E, Desjardins CD, Rohde P. Young women who develop anorexia nervosa exhibit a persistently low premorbid body weight on average: A longitudinal investigation of an important etiologic clue. J Psychopathol Clin Sci. 2022 Jul;131(5):479-492. doi: 10.1037/abn0000762. Epub 2022 Jun 2. PMID 35653756
- [Derived] Akers L, Rohde P, Shaw H, Stice E. Cost-Effectiveness Comparison of Delivery Modalities for a Dissonance-Based Eating Disorder Prevention Program over 4-Year Follow-Up. Prev Sci. 2021 Nov;22(8):1086-1095. doi: 10.1007/s11121-021-01264-1. Epub 2021 Jun 21. PMID 34152570
- [Derived] Stice E, Rohde P, Shaw H, Desjardins C. Weight suppression increases odds for future onset of anorexia nervosa, bulimia nervosa, and purging disorder, but not binge eating disorder. Am J Clin Nutr. 2020 Oct 1;112(4):941-947. doi: 10.1093/ajcn/nqaa146. PMID 32534455
- [Derived] Stice E, Rohde P, Shaw H, Gau JM. Clinician-led, peer-led, and internet-delivered dissonance-based eating disorder prevention programs: Effectiveness of these delivery modalities through 4-year follow-up. J Consult Clin Psychol. 2020 May;88(5):481-494. doi: 10.1037/ccp0000493. Epub 2020 Feb 24. PMID 32091226
- [Derived] Stice E, Rohde P, Shaw H, Gau JM. Clinician-led, peer-led, and internet-delivered dissonance-based eating disorder prevention programs: Acute effectiveness of these delivery modalities. J Consult Clin Psychol. 2017 Sep;85(9):883-895. doi: 10.1037/ccp0000211. Epub 2017 Apr 20. PMID 28425735